CLINICAL TRIAL: NCT07038356
Title: Effects of Continued Administration of Empagliflozin in Patients With Heart Failure on Active SGLT2 Inhibitor Treatment Admitted for Acute Decompensated Heart Failure
Acronym: EMPA-CON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Christian Schulze (Other)
Responsible Party: Sponsor-Investigator, Christian Schulze, Director of Department of Internal Medicine I at Jena University Hospital and Professor of Medicine at Friedrich Schiller University Jena, Jena University Hospital
Organization: Jena University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMPA-CON_ZKSJ0162; 2024-517977-26-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-23; First posted 2025-06-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Acute Decompensated Heart Failure (ADHF)
MeSH Terms: interventions — empagliflozin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): Randomized treatment with placebo (one tablet) daily from day 1 until the day of hospital discharge, but no longer than 30 days, followed by 10 mg empagliflozin (Jardiance, one tablet) daily until day 90.
  Interventions: Drug: Placebo
- intervention (Active Comparator): Drug: Empagliflozin (10 mg/day), film-coated tablet Randomized treatment with 10 mg empagliflozin (Jardiance, one tablet) or placebo daily from day 1 until the day of hospital discharge, but no longer than 30 days, followed by 10 mg empagliflozin (Jardiance, one tablet) daily until day 90
  Interventions: Drug: Empagliflozin 10 MG Oral Tablet [Jardiance]

INTERVENTIONS:
Drug: Empagliflozin 10 MG Oral Tablet [Jardiance] — Randomized treatment with 10 mg empagliflozin (Jardiance, one tablet) daily from day 1 until the day of hospital discharge, but no longer than 30 days, followed by 10 mg empagliflozin (Jardiance, one tablet) daily until day 90
  Arms: intervention
Drug: Placebo — Randomized treatment with placebo (one tablet) daily from day 1 until the day of hospital discharge, but no longer than 30 days, followed by 10 mg empagliflozin (Jardiance, one tablet) daily until day 90
  Arms: control

SUMMARY:
The goal of this clinical trial is to test the hypothesis that the continuation of empagliflozin during decongestive therapy in the setting of acute decompensated and hospitalized heart failure patients is not inferior compared to therapy cessation during the acute heart failure hospitalization.

Randomized treatment (plus standard medical care) in patients with acute decompensated heart failure is one (1) tablet daily of empagliflozin 10 mg or matching placebo during the in-hospital stay (up to a maximum of 30 days), followed by treatment with empagliflozin 10 mg daily after discharge (but no later than day 31) until day 90.

The primary outcome measure is the combined hierarchical endpoint of all-cause mortality, heart failure hospitalization and worsening renal function at 90 days after admission.

Secondary outcome measures are the effects on urine output, diuretic efficiency, quality-of-life and the need for further administration of diuretics.

Participants will

* Take one tablet of study medication once daily (day 1 to day 90)
* Restrict fluid intake to 1.5 liters of fluid per day and record the daily fluid intake for the study from day 1 to day 6 in the patient diary
* Measure the urine output (day 1 to day 6)
* Fill in Questionnaires (EQ-5D-3L (3-level version of the EuroQol five dimensional descriptive system), KCCQ-12 (Kansas City Cardiomyopathy Questionnaire comprising 12 items)) on day 0 (Baseline), at hospital discharge, and on day 30

ELIGIBILITY:
Inclusion Criteria:

* Patients (age ≥ 18 years) with acute decompensated heart failure (HF) according to clinical assessment on active therapy with a SGLT2 inhibitor
* Brain Natriuretic Peptide (BNP) >100 pg/ml or N-terminal pro-BNP (NTproBNP) >300 pg/ml
* Written informed consent obtained
* Women of childbearing potential: negative pregnancy test and use of a highly effective method of contraception

Exclusion Criteria:

* Type 1 diabetes mellitus
* Chronic Kidney Disease (CKD) with eGFR<20 ml/min, or end-stage renal failure with the need for chronic dialysis treatment
* Acute kidney injury (AKI) requiring dialysis treatment
* Known intolerance to empagliflozin
* Acute heart failure without signs of congestion ("dry" patient)
* Indication for coronary angiography or any foreseeable administration of a contrast media
* Need for hemofiltration or any other form of extracorporeal therapy
* Planned surgery
* Previous participation in this trial or recent participation in another clinical trial (within the last 4 weeks before inclusion)
* Identification of any causes of heart failure leading to decompensation that needs urgent management (like acute coronary syndrome, severe unstable arrhythmias, mechanical causes, acute pulmonary embolism)
* Incapacity to understand and / or to provide written informed consent
* Obvious uncontrolled substance abuse
* Pregnancy, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Four-step hierarchical composite primary endpoint; win ratio based on the following parameters (day 90): time to all-cause death, number of heart failure events per patient, time to first heart failure event, eGFR decrease from baseline to day 90 | day 90
  The study uses a four-step hierarchical composite primary endpoint (win ratio):
  1. time to all-cause death, days (day 90)
  2. number of heart failure events per patient (day 90)
  3. time to first heart failure event, days (day 90)
  4. eGFR decrease from baseline to day 90 (with a between-patient threshold defined as ≥5 ml/min/1.73 m²)

SECONDARY OUTCOMES:
Cardiovascular and total mortality on day 90 | day 90
Number of patients alive and without re-hospitalization on day 90 | day 90
Re-hospitalization after initial discharge, including reason: time to first rehospitalization after discharge | day 90
Re-hospitalization after initial discharge, including reason: numbers of re-hospitalizations | day 90
Number of patients with a decrease in eGFR of 5 ml/min/1.73 m² or more from baseline to day 90 | day 90
Daily and cumulative urine output (UOP, ml) measured from day 1 until day 6 | day 1 until day 6
Diuretic efficiency (ml urine per mg furosemide equivalent) from day 1 to day 6 | day 1 until day 6
Change in body weight from baseline to day 1, day 3, day 6, discharge (supposed between day 6-10), day 30, and day 90 | day 1, day 3, day 6, discharge (supposed between day 6-10), day 30, and day 90
Renal function at baseline, day 3, day 6, day 30, and day 90 | baseline, day 3, day 6, day 30, and day 90
  * Decrease in eGFR of >20 ml/min/1.73 m2
  * Doubling of serum creatinine
  * Need for renal replacement therapy
  * Total urinary sodium excretion and fractional excretion of sodium
Liver function: bilirubin (nmol/ml) at baseline, day 3, day 6, day 30, and day 90 | baseline, day 3, day 6, day 30, and day 90
Liver function: serum aminotransferases (µmol/l*s) at baseline, day 3, day 6, day 30, and day 90 | baseline, day 3, day 6, day 30, and day 90
Liver function: relevant change in coagulation status (Quick/INR, %, 3X upper limit of normal) at baseline, day 3, day 6, day 30, and day 90 | baseline, day 3, day 6, day 30, and day 90
Change in NT-proBNP (N-terminal pro Brain natriuretic peptide, pg/ml) (alternatively calculated from BNP, Brain natriuretic peptide, pg/ml) from baseline to day 6, day 30, and day 90 | baseline to day 6, day 30, and day 90
Quality of life (EQ-5D-3L questionnaire, 3-level version of the EuroQol five dimensional descriptive system ) on day 0, at hospital discharge (supposed between day 6-10), and on day 30 | day 0, at hospital discharge (supposed between day 6-10), and on day 30
  Quality of life: EQ-5D-3L questionaire. The EQ-5D-3L questionnaire consists of two parts: part one contains questions about patients mobility, self-care, usual activities, pain/discomfort, anxiety/depression, with scores from 1 (no problem), 2 (some problems), and 3 (extreme problems). Part two measures patients health on a scale from 0 (the worst imaginable health) to 100 (the best imaginable health), on day 0, at hospital discharge (supposed between day 6-10), and on day 30
Severity of heart failure (HF): KCCQ-12 questionnaire (Kansas City Cardiomyopathy Questionnaire comprising 12 items) on day 0, at hospital discharge (supposed between day 6-10), and on day 30 | day 0, at hospital discharge (supposed between day 6-10), and on day 30
  KCCQ-12 questionnaire: scores range from 0 to 100, with higher scores indicating better health status, on day 0, at hospital discharge (supposed between day 6-10), and on day 30
Intermediate Care Unit (IMC) / Intensive Care Unit (ICU) and hospital length of stay, days until discharge (supposed between day 6-10) | discharge (supposed between day 6-10)
Single parameters of primary endpoint: time to all-cause death (day 90) | day 90
Single parameters of primary endpoint: number of heart failure events per patient (day 90) | day 90
Single parameters of primary endpoint: time to first heart failure event (day 90) | day 90
Single parameters of primary endpoint: eGFR decrease from baseline to day 90 (ml/min/1.73 m²) | day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Jena University Hospital, Jena, Thuringia, Germany